CLINICAL TRIAL: NCT06842537
Title: A Phase I Clinical Trial to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of SYH2062 Injection in Healthy Chinese Volunteers
Brief Title: Study of SYH2062 Injection in Healthy Chinese Volunteers
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: CSPC Zhongnuo Pharmaceutical (Shijiazhuang) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SYH2062-001
Record Dates: First submitted 2025-02-19; First posted 2025-02-24 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-02

CONDITIONS: Healthy Chinese Volunteers

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SYH2062 injection (Experimental)
  Interventions: Drug: SYH2062 injection
- SYH2062-Matching placebo (Placebo Comparator)
  Interventions: Drug: SYH2062-Matching placebo

INTERVENTIONS:
Drug: SYH2062 injection — SYH2062 for sc injection
  Arms: SYH2062 injection
Drug: SYH2062-Matching placebo — Normal saline matching volume of SYH2062 doses will be administered
  Arms: SYH2062-Matching placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, efficacy, pharmacodynamics and pharmacokinetics of SYH2062 injection in healthy Chinese volunteers

DETAILED DESCRIPTION:
A Phase 1, randomized, double-Blind, placebo-Controlled study to evaluate the safety, tolerability, pharmacokinetic and pharmacodynamic characteristics of SYH2062 injection after a single administration in healthy subjects

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must give informed consent before the trial, fully understand the content, process and possible adverse reactions, and voluntarily sign a written informed consent.
2. Age of 18 - 55 years (inclusive).
3. BMI: 19.0-26.0 kg/m^2 (inclusive), with a minimum weight of 50 kg (inclusive) for males and 45 kg (inclusive) for females.
4. Has Systolic blood pressure (SBP) ≥100 mmHg and <140 mmHg and diastolic blood pressure (DBP) ≥60 mmHg and <90 mmHg at screening;
5. The subjects can communicate well with the investigators and complete the trial according to protocol.

Exclusion Criteria:

Allergic constitution, or known history of allergy to the components of the study drug or similar drugs.

2 Subjects with the following diseases of clinical significance (including but not limited to diseases of the circulatory system, diseases of the blood or hematopoietic system, diseases of the respiratory system, diseases of the endocrine system, diseases of the urinary system, diseases of the digestive system, neurological or mental diseases, infections, tumors, serious injuries).

3 Those who underwent major surgery within 6 months prior to initial administration, or who planned to undergo surgery during the study.

4 Blood loss or blood donation of more than 200 mL within 3 months prior to initial administration (except for female menstrual period), and/or platelet donation within 2 weeks prior to initial administration.

5 Positive urine drug screening. 6 Those who smoked more than 5 cigarettes per day within 3 months prior to screening and/or did not agree to refrain from using any tobacco products during hospitalization.

7 Regular drinkers within 6 months prior to screening, i.e., those who drank more than 14 units of alcohol per week, and/or those who could not stop drinking alcohol during their hospitalization, and/or test positive for breath alcohol.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) | up to approximately 12 months

SECONDARY OUTCOMES:
Change from Baseline in Blood Angiotensinogen (AGT) Level | up to approximately 12 months
Change from Baseline in in plasma renin concentration | up to approximately 12 months
Change from Baseline in in plasma renin activity | up to approximately 12 months
Change from Baseline in in angiotensin I | up to approximately 12 months
Change from Baseline in in angiotensin II | up to approximately 12 months
Change from Baseline in in plasma aldosterone | up to approximately 12 months
To characterize the Cmax of single dose of SYH2062 | Up to Day 3
To characterize the AUC of single dose of SYH2062 | Up to Day 3
Number of Participants With Anti- SYH2062 Antibodies | up to approximately 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese Academy of Medical Science and Peking Union Medical College Hospital, Beijing, Beijing Municipality, China